CLINICAL TRIAL: NCT05908461
Title: The Early Childhood Friendship Project: Testing Key Mechanisms and the Moderating Role of Physiological Reactivity
Brief Title: The Early Childhood Friendship Project - Phase 3
Acronym: ECFP-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jamie M. Ostrov, Ph.D., Professor of Psychology, Clinical Area Head, Director of Clinical Training, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00004375; 1R01HD105496-01A1 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive the Early Childhood Friendship project intervention (8x10-min puppet shows, 7x5-min gross motor activities7x5-min passive activities, up to 3x1-hour in-vivo behavioral reinforcement periods).
  Interventions: Behavioral: Early Childhood Friendship Project
- Control Group (No Intervention): Participants will not receive the Early Childhood Friendship project intervention.

INTERVENTIONS:
Behavioral: Early Childhood Friendship Project — Classroom-based intervention where teachers will implement 8 10-minute puppet shows, 7 5-minute active gross motor activities to reinforce the social skill of the week, and 7 5-minute passive rehearsal activities such as making their own puppet and practicing the steps of the week. Up to three 1 hour in vivo behavioral reinforcement periods will occur per week and during these free play sessions teachers and the main puppet will use developmentally appropriate praise to reinforce the use of the social skills of the week.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess the impact of the Early Childhood Friendship Project (ECFP) on changes in aggression/peer victimization subtypes, prosocial behavior, and social and academic competence with a teacher-implemented (with coaching) version of the program. Further, investigators will examine whether changes in executive functioning, emotion regulation, and hostile attribution biases indirectly account for the program effects. Investigators will test if physiological reactivity (skin conductance and respiratory sinus arrhythmia) serves as moderators of intervention effects. Data will be collected from 600 children (30 randomly assigned preschool classrooms) diverse in socioeconomic status and race/ethnicity. Investigators will use multiple methods (school-based observations, direct academic assessments, child interviews, physiological reactivity using two tasks, observer, caregiver, and teacher reports) to assess the efficacy of the program, hypothesized mechanisms, and role of physiology as a moderator of intervention effects. The duration of the effects will be tested at both 4 month and 12-month follow-up and will thus demonstrate the impact the program has on children's school readiness and transition to kindergarten. It is expected that preschool children randomly assigned to the ECFP intervention relative to the control condition will show significant and moderate reductions in physical and relational aggression/victimization at post-test and follow-up; the ECFP intervention group will also show increases in prosocial behavior, social competence, and academic competence, relative to the control group at post-test and follow-up (4-months at the end of preschool and 12 months after transitioning to kindergarten). Additionally, it is hypothesized that changes in executive functioning, emotion regulation, and hostile attribution biases will mediate treatment effects from baseline to respective follow-ups. It is anticipated that these hypothesis will be moderated by gender such that effects will be stronger for girls relative to boys. Finally, it is hypothesized that physiological reactivity will act as a moderator of intervention effects and of the executive functioning, emotion regulation, and hostile attribution biases mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* A child is eligible if attending one of the participating child care centers in the greater Buffalo region of Western New York and planning to enter kindergarten in the fall.

Exclusion Criteria:

* None

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2027-04-16 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Observations of Physical Aggression (Early Childhood Observation System - Frequency Count up to 8 Sampling Sessions) | Up to 12 weeks post-intervention completion.
  Physical aggression will be assessed via focal child sampling with continuous recording observation for each participating child. Each observation is 10 minutes for up to 8 separate observations (i.e., frequency counts divided by number of sessions out of 8 sessions).
Observations of Prosocial Behavior (Early Childhood Observation System - Frequency Count up to 8 Sampling Sessions) | Up to 12 weeks post-intervention completion.
  Prosocial behavior will be assessed via focal child sampling with continuous recording observations for each participating child. Each observation is 10 minutes for up to 8 separate observations (i.e., frequency counts divided by number of sessions out of 8 sessions).
Observations of Relational Aggression (Early Childhood Observation System - Frequency Count up to 8 Sampling Sessions) | Up to 12 weeks post-intervention completion.
  Relational aggression will be assessed via focal child sampling with continuous recording observations for each participating child. Each observation is 10 minutes for up to 8 separate observations (i.e., frequency counts divided by number of sessions out of 8 sessions).
Observations of Physical Victimization (Early Childhood Observation System - Frequency Count up to 8 Sampling Sessions) | Up to 12 weeks post-intervention completion.
  Physical victimization will be assessed via focal child sampling with continuous recording observations for each participating child. Each observation is 10 minutes for up to 8 separate observations (i.e., frequency counts divided by number of sessions out of 8 sessions).
Observations of Relational Victimization (Early Childhood Observation System - Frequency Count up to 8 Sampling Sessions) | Up to 12 weeks post-intervention completion.
  Relational victimization will be assessed via focal child sampling with continuous recording observations for each participating child. Each observation is 10 minutes for up to 8 separate observations (i.e., frequency counts divided by number of sessions out of 8 sessions).
Dynamic Indicators of Basic Early Learning (DIBELS) - Sound Fluency | Up to 4 months post-intervention completion.
  Sound fluency will be measured using the DIBELS - Sound Fluency measure. Scores are calculated as the correct initial sounds per minute, with higher scores indicating greater performance on this measure.
Dynamic Indicators of Basic Early Learning (DIBELS) - Letter Naming Fluency | Up to 4 months post-intervention completion.
  Letter naming fluency will be measured using the DIBELS - Letter Naming Fluency measure. Scores on this measure range from 0 to 110, with higher scores indicating greater performance.
Early Numeracy Skills: Set Comparison | Up to 4 months post-intervention completion.
  Early numeracy will be assessed using the task set comparisons. In this activity, a child is presented with four sets of dots representing different amounts and asked which has the most or fewest dots. A child's score is a sum of correct responses. Scores range from 0-6, with higher scores indicating stronger performance.
Early Numeracy Skills: One-to-One Counting | Up to 4 months post-intervention completion.
  Early numeracy will be assessed using the task one-to-one counting. In this task, a child is presented with a set of dots and asked to count the set. A child's score is sum of correct responses. Scores range from 0 to 5, with higher scores indicating stronger performance.
Early Numeracy Skills: Verbal Counting | Up to 4 months post-intervention completion.
  Early numeracy will be assessed using the task verbal counting. In this task, a child is asked to count as high as possible until the child makes a mistake or correctly counts up to 100. A child's score is a single score based on correct counting out of 100. Scores range from 1-7, with higher scores indicating stronger performance.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Relational Victimization Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the PPVM-T-R Relational Victimization subscale to assess relational victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of relational victimization.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Physical Victimization Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the PPVM-T-R physical victimization subscale to assess physical victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical victimization.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Physical Victimization Subscale | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete the PPVM-T-R physical victimization subscale to assess physical victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical victimization.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Relational Victimization Subscale | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete the PPVM-T-R relational aggression subscale to assess relational victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical victimization.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Physical Victimization Subscale | Up to 4 months post-intervention completion.
  Research assistant observers will complete the PPVM-T-R physical victimization to assess physical victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical victimization.
Preschool Peer Victimization Measure - Teacher Report - Revised (PPVM-T-R): Relational Victimization Subscale | Up to 4 months post-intervention completion.
  Research assistant observers will complete the PPVM-T-R relational victimization subscale to assess relational victimization. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical victimization.
Preschool Social Behavior Scale - Teacher Report (PSBS-TR): Physical Aggression Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the PSBS-TR physical aggression subscale to assess physical aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Relational Aggression Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the PSBS-TR relational aggression subscale to assess relational aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of relational aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Prosocial Behavior Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the PSBS-TR prosocial behavior subscale to assess prosocial behavior. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of prosocial behavior.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Relational Aggression Subscale | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete the PSBS-TR relational aggression subscale to assess relational aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of relational aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Physical Aggression Subscale | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete the PSBS-TR physical aggression subscale to assess physical aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Prosocial Behavior Subscale | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete the PSBS-TR prosocial behavior subscale to assess prosocial behavior. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Physical Aggression Subscale | Up to 4 months post-intervention completion.
  Research assistant observers will complete the PSBS-TR physical aggression subscale to assess physical aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Relational Aggression Subscale | Up to 4 months post-intervention completion.
  Research assistant observers will complete the PSBS-TR relational aggression subscale to assess relational aggression. Raw scores are 6-30 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of relational aggression.
Preschool Social Behavioral Scale - Teacher Report (PSBS-TR): Prosocial Behavior Subscale | Up to 4 months post-intervention completion.
  Research assistant observers will complete the PSBS-TR prosocial behavior subscale to assess prosocial behavior. Raw scores are 4-20 with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of physical aggression.
MacArthur Health and Behavior Questionnaire (HBQ) - School Performance Subscale | Up to 12 weeks post-intervention completion.
  Teachers will complete the HBQ school performance subscale to assess academic competence. Raw scores range from 5-25 with average scores on this measure ranging from 1-5, and with higher scores indicate higher levels of academic competence.
MacArthur Health and Behavior Questionnaire (HBQ) - School Performance Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the HBQ school performance subscale to assess academic competence. Raw scores range from 5-25, with average scores on this measure ranging from 1-5, and with higher scores indicating higher levels of academic competence.
MacArthur Health and Behavior Questionnaire (HBQ) - School Engagement Subscale | Up to 12 weeks post-intervention completion.
  Teachers will complete the HBQ school engagement subscale to assess school engagement. Raw scores range from 0-16, with average scores on this measure ranging from 0-2, and with higher scores indicating higher levels of school engagement.
MacArthur Health and Behavior Questionnaire (HBQ) - School Engagement Subscale | An average of 12 months post-intervention completion.
  Teachers will complete the HBQ school engagement subscale to assess school engagement. Raw scores range from 0-16, with average scores on this measure ranging from 0-2, and with higher scores indicating higher levels of school engagement.
Social Skills Rating Scale (SSRS) | An average of 12 months post-intervention completion.
  Teachers will complete this standard measure of social skills. Raw scores range from 0 to 60, with average scores on this measure ranging from 0-2, and with higher scores indicating higher levels of social skills.
Social Skills Rating Scale (SSRS) | Up to 12 weeks post-intervention completion.
  Research assistant observers will complete this standard measure of social skills. Raw scores range from 0 to 60, with average scores on this measure ranging from 0-2, and with higher scores indicating higher levels of social skills.
Social Skills Rating Scale (SSRS) | Up to 4 months post-intervention completion.
  Research assistant observers will complete this standard measure of social skills. Raw scores range from 0 to 60, with average scores on this measure ranging from 0-2, and with higher scores indicating higher levels of social skills.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Ostrov, Ph.D., Principal Investigator — University at Buffalo, SUNY
Locations (1):
- University at Buffalo, SUNY, Buffalo, New York, United States